CLINICAL TRIAL: NCT05849922
Title: A Randomized, Double-blind, Placebo-controlled, Proof-of-concept Study Assessing the Efficacy and Safety of an Anti-TNF-OX40L NANOBODY® Molecule, SAR442970, in Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Test the Efficacy and Safety of SAR442970 in Adults With Hidradenitis Suppurativa
Acronym: HS OBTAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT16852; U1111-1280-6493 (Registry Identifier: ICTRP); 2022-502370-17 (Registry Identifier: CTIS); 2022-502370-17 (EudraCT Number)
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR442970 (Experimental): Participants received SAR442970 once every two weeks (Q2W) in Period A (Day 1 to Week 16). Participants received SAR442970 Q2W in Period B (Up to Week 28).
  Interventions: Drug: SAR442970
- Placebo (Placebo Comparator): Participants received placebo Q2W in Period A (Day 1 to Week 16). Participants received SAR442970 Q2W in Period B (Up to Week 28).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR442970 — 1 mL extractable volume of 150 mg/mL SAR442970 filled in 2 mL glass vial
  Arms: SAR442970
Drug: Placebo — 1 mL extractable volume of placebo filled in 2 mL glass vial
  Arms: Placebo

SUMMARY:
This was a Phase 2 study in adult participants with moderate to severe hidradenitis suppurativa (HS). The purpose of the study was to evaluate the efficacy and safety of SAR442970 compared to placebo.

DETAILED DESCRIPTION:
The study duration was up to 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a history of signs and symptoms consistent with hidradenitis suppurativa (HS) for at least 1 year prior to Baseline.
* Participants had to have HS lesions present in at least 2 distinct anatomic areas (eg, left and right axilla; or left axilla and left inguinocrural fold), one of which had to be Hurley Stage II or Hurley Stage III.
* Participant had to have had an inadequate response to a trial of an oral antibiotic for treatment of HS, exhibited recurrence after discontinuation of antibiotics, demonstrated intolerance to antibiotics, or had a contraindication to oral antibiotics for treatment of their HS as assessed by the Investigator through participant interview and review of medical history.
* Participants had to be either biologic and small molecule immunosuppressive-naïve or TNF-experienced.
* Participant had to have a total abscess and inflammatory nodule (AN) count of ≥3 at the Baseline visit.
* Participant had to have a draining tunnel count of ≤20 at the Baseline visit.
* Participant had to have a C-reactive protein (CRP) >3 mg/L at the screening visit.
* Participant who was a candidate for systemic treatment per Investigator's judgment.

Exclusion Criteria:

* Any other active skin disease or condition (eg, bacterial, fungal or viral infection) that might have interfered with assessment of HS
* History of recurrent or recent serious infection
* Known history of or suspected significant current immunosuppression
* History of solid organ transplant
* History of splenectomy
* History of moderate to severe congestive heart failure
* Receipt of a live vaccine 12 week prior to Baseline visit or receipt of a killed vaccine 2 weeks prior to Baseline visit
* History of demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease
* Participants with a history of malignancy or lymphoproliferative disease other than adequately treated or nonmetastatic squamous cell carcinoma, or nonmetastatic basal cell carcinoma of the skin that was excised and completely cured
* Participants with a diagnosis of inflammatory conditions other than HS
* Presence of active suicidal ideation, or positive suicide behavior or participant had a lifetime history of suicide attempt, or participant had had suicidal ideation in the past 6 months as indicated by a positive response using the screening or Baseline version of the Columbia-Suicide Severity Rating Scale (C-SSRS) or as assessed by the Investigator through participant interview and review of medical history
* A history of an adverse event (AE) to anti-TNF therapy (examples included, but were not limited, to serum sickness or anaphylaxis) for an HS or non-HS indication that would contraindicate readministration of an anti-TNF class therapy
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicated participation in the study
* Female participants who were breastfeeding or considering becoming pregnant during the study
* History (within last 2 years prior to Baseline) of prescription drug or substance abuse, including alcohol, considered significant by the Investigator
* Laboratory exclusion criteria applied.

The above information was not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2025-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (45):
- United States (6):
  - Medical Dermatology Specialists Site Number : 8400007, Phoenix, Arizona
  - Renstar Medical Research Site Number : 8400011, Ocala, Florida
  - ForCare Clinical Research Site Number : 8400006, Tampa, Florida
  - Advanced Medical Research PC Site Number : 8400002, Sandy Springs, Georgia
  - Clinical Partners, LLC Site Number : 8400010, Johnston, Rhode Island
  - Center for Clinical Studies, LTD. LLP Site Number : 8400003, Houston, Texas
- Australia (2):
  - Investigational Site Number : 0360002, Liverpool, New South Wales
  - Investigational Site Number : 0360003, Woolloongabba, Queensland
- Investigational Site Number : 0560001, Leuven, Belgium
- Canada (4):
  - Investigational Site Number : 1240001, Barrie, Ontario
  - Investigational Site Number : 1240002, London, Ontario
  - Investigational Site Number : 1240004, Newmarket, Ontario
  - Investigational Site Number : 1240007, Québec
- Chile (3):
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
- Czechia (3):
  - Investigational Site Number : 2030003, Ostrava - Poruba
  - Investigational Site Number : 2030001, Prague
  - Investigational Site Number : 2030002, Praha 5 - Motol
- Investigational Site Number : 2080001, Roskilde, Denmark
- France (3):
  - Investigational Site Number : 2500001, Lyon
  - Investigational Site Number : 2500002, Nice
  - Investigational Site Number : 2500003, Reims
- Germany (5):
  - Investigational Site Number : 2760005, Berlin
  - Investigational Site Number : 2760008, Bochum
  - Investigational Site Number : 2760002, Frankfurt am Main
  - Investigational Site Number : 2760004, Mainz
  - Investigational Site Number : 2760001, Münster
- Greece (2):
  - Investigational Site Number : 3000003, Athens
  - Investigational Site Number : 3000001, Athens
- Italy (3):
  - Investigational Site Number : 3800001, Milan, Lombardy
  - Investigational Site Number : 3800002, Rozzano, Lombardy
  - Investigational Site Number : 3800003, Catania
- Netherlands (2):
  - Investigational Site Number : 5280001, Groningen
  - Investigational Site Number : 5280003, Rotterdam
- Poland (4):
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160004, Lodz
  - Investigational Site Number : 6160003, Wroclaw
  - Investigational Site Number : 6160002, Wroclaw
- Spain (5):
  - Investigational Site Number : 7240003, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240006, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240001, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240004, Manises, Valencia
  - Investigational Site Number : 7240005, Córdoba
- Investigational Site Number : 7520001, Älvsjö, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Lin J, Radhakrishnan J. What Are Baskets, Umbrellas, and Platforms Doing in Nephrology Clinical Trials? J Am Soc Nephrol. 2025 Feb 3;36(8):1652-1654. doi: 10.1681/ASN.0000000648. No abstract available. PMID 39899371
- See also: ACT16852 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25201&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to screen participants in June 2023 and concluded enrollment in April 2024.
Pre-assignment Details: A total of 86 participants were randomized in a 2:1 ratio to receive either SAR442970 150 milligrams (mg) or a matching placebo. The study consisted of a screening period (up to 4 weeks), a treatment period (16-week Period A [double blind {DB}] and 12-week Period B [open-label extension {OLE}]), and safety follow-up period (8 weeks).
Groups:
- Period A: Placebo: Participants received SAR442970 matched placebo every 2 weeks (Q2W) via subcutaneous (SC) injection from Day 1 to Week 16 in Period A (DB period).
- Period A: SAR442970: Participants received SAR442970 150 mg Q2W via SC injection from Day 1 to Week 16 in Period A (DB period).
- Period B: Placebo-SAR442970: Participants who received SAR442970 matched placebo in Period A (DB period) received SAR442970 150 mg Q2W via SC injection from Week 16 to Week 28 in Period B (OLE period).
- Period B: SAR442970-SAR442970: Participants who received SAR442970 in Period A (DB period) received SAR442970 150 mg Q2W via SC injection from Week 16 to Week 28 in Period B (OLE period).
Period: Period A (DB): Up to Week 16
Arm/Group | Period A: Placebo | Period A: SAR442970 | Period B: Placebo-SAR442970 | Period B: SAR442970-SAR442970
Started | 28 (Note: Reason for not completed = Reason for permanent study drug discontinuation.) | 58 (Note: Reason for not completed = Reason for permanent study drug discontinuation.) | 0 | 0
Completed | 26 | 52 | 0 | 0
Not Completed | 2 | 6 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Other | 1 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Period: Period B (OLE): From Week 16 to Week 28
Arm/Group | Period A: Placebo | Period A: SAR442970 | Period B: Placebo-SAR442970 | Period B: SAR442970-SAR442970
Started | 0 | 0 | 26 (Eligible participants who completed the Period A (DB period) entered Period B (OLE period). Note: Reason for not completed = Reason for permanent study drug discontinuation.) | 51 (1 participant completed the Period A (DB period) but did not enroll into the Period B (OLE period). As a result, 52 participants completed Period A, but only 51 participants entered Period B. Note: Reason for not completed = Reason for permanent study drug discontinuation.)
Completed | 0 | 0 | 24 | 45
Not Completed | 0 | 0 | 2 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Non-compliance with study schedule | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Other | 0 | 0 | 0 | 2
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The randomized population included all participants from screened population who were allocated to a randomized study drug by interactive response technology regardless of whether the study drug was received or not.
Groups:
- Period A: Placebo: Participants received SAR442970 matched placebo Q2W via SC injection from Day 1 to Week 16 in Period A (DB period).
- Total: Total of all reporting groups
Arm/Group | Period A: Placebo | Period A: SAR442970 | Total
Number analyzed (Participants) | 28 | 58 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (13.2) | 36.3 (12.2) | 36.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 38 | 53
  Male | 13 | 20 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 16 | 50 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Period A (DB Period): Percentage of Biologic and Small Molecule Immunosuppressive-Naïve Participants Who Achieved Hidradenitis Suppurativa Clinical Response (HiSCR50) at Week 16
Description: The HiSCR50 was used for assessing HS treatment effectiveness in controlling inflammatory manifestations in the population. HiSCR50 was defined as >=50% reduction from baseline in the total abscess and inflammatory nodule (AN) count, with no increase from baseline in abscess or draining tunnel count. Baseline was defined as the last available value before the first dose of DB study drug. Percentages are rounded off to the tenth decimal place.
Time Frame: Week 16
Population: The biologic and small molecule immunosuppressive-naïve population included all randomized participants in the biologic and small molecule immunosuppressive-naïve subgroup who had taken at least 1 dose of study drug during Period A.
Measure: Number; unit: percentage of participants
Arm/Group | Period A: Placebo | Period A: SAR442970
Number analyzed (Participants) | 23 | 48
percentage of participants | 39.1 | 66.7
Statistical Analysis 1: Comparison: Period A: Placebo vs Period A: SAR442970; Bayesian logistic regression approach was done. Here, RR=response rate; Test type: Other; Median posterior RR difference = 29, 90% CI 2-sided [10 to 47]
Statistical Analysis 2: Comparison: Period A: Placebo vs Period A: SAR442970; Bayesian logistic regression approach was done. Here, Pr=posterior probability of superiority; Test type: Other; Pr[Diff > 0%](%) = 99.3

2. Secondary Outcome: Period A (DB Period): Time to Onset of Achieving Hidradenitis Suppurativa Clinical Response (HiSCR50)
Description: Time to onset of achieving HiSCR50 during the DB period was defined as the time from randomization to the first time of achieving HiSCR50 by Week 16. HiSCR50 was defined as >=50% reduction from baseline in the total AN count, with no increase from baseline in abscess or draining tunnel count. Baseline was defined as the last available value before the first dose of DB study drug.
Time Frame: Up to Week 16
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Period A: Placebo | Period A: SAR442970
Number analyzed (Participants) | 23 | 48
days | 113.00 [29.000 to NA] — NA indicates that the upper limit of the 90% confidence interval was not estimable due to insufficient number of participants achieving HiSCR50 by the end of the DB period. | 29.00 [17.000 to 29.000]

3. Secondary Outcome: Period A (DB Period): Percentage of Participants Who Achieved Hidradenitis Suppurativa Clinical Response (HiSCR75) at Week 16
Description: The HiSCR75 was used for assessing HS treatment effectiveness in controlling inflammatory manifestations in the population. HiSCR75 was defined as >=75% reduction from baseline in the total AN count, with no increase from baseline in abscess or draining tunnel count. Baseline was defined as the last available value before the first dose of DB study drug.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Period A: Placebo | Period A: SAR442970
Number analyzed (Participants) | 23 | 48
percentage of participants | 21.7 | 54.2

4. Secondary Outcome: Period A (DB Period): Percentage of Participants Who Achieved Hidradenitis Suppurativa Clinical Response (HiSCR90) at Week 16
Description: The HiSCR90 was used for assessing HS treatment effectiveness in controlling inflammatory manifestations in the population. HiSCR90 was defined as >=90% reduction from baseline in the total AN count, with no increase from baseline in abscess or draining tunnel count. Baseline was defined as the last available value before the first dose of DB study drug.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Period A: Placebo | Period A: SAR442970
Number analyzed (Participants) | 23 | 48
percentage of participants | 8.7 | 31.3

5. Secondary Outcome: Period A (DB Period): Percentage of Participants Who Experienced Improvement by at Least 1 International Hidradenitis Suppurativa Severity Score System (IHS4) Stage at Week 16
Description: The IHS4 was a validated tool to assess HS severity. The determination of IHS4 required counting inflammatory nodules, abscesses and draining tunnels and multiplying each by a specific coefficient. IHS4 score was calculated as: (number of inflammatory nodules multiplied by 1) + (number of abscesses multiplied by 2) + (number of draining tunnels multiplied by 4). A categorial IHS4 score was derived from this weighted score with total score range: mild: (<=3), moderate: (4 to 10) and severe: (>=11); higher scores indicated worse outcomes. Improvement in IHS4 by >=1 IHS4 stage was considered clinically meaningful.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Period A: Placebo | Period A: SAR442970
Number analyzed (Participants) | 23 | 48
percentage of participants | 56.5 | 83.3

6. Secondary Outcome: Period A (DB Period): Change From Baseline at Week 16 in Absolute Score in International Hidradenitis Suppurativa Severity Score System (IHS4)
Description: The IHS4 was a validated tool to assess HS severity. The determination of IHS4 required counting inflammatory nodules, abscesses and draining tunnels and multiplying each by a specific coefficient. IHS4 score was calculated as: (number of inflammatory nodules multiplied by 1) + (number of abscesses multiplied by 2) + (number of draining tunnels multiplied by 4). A categorial IHS4 score was derived from this weighted score with total score range: mild: (<=3), moderate: (4 to 10) and severe: (>=11); higher scores indicated worse outcomes. Baseline was defined as the last available value before the first dose of DB study drug.
Time Frame: Baseline (Day 1) and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Period A: Placebo | Period A: SAR442970
Number analyzed (Participants) | 23 | 48
score on a scale | -7.3 (19.5) | -18.1 (18.6)

7. Secondary Outcome: Period A (DB Period): Percentage of Participants Who Experienced a Flare Relative to Baseline at Week 16
Description: HS flare was defined as >=25% increase in AN count with a >=2 increase from baseline by Week 16. Baseline was defined as the last available value before the first dose of DB study drug.
Time Frame: Baseline (Day 1) and Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Period A: Placebo | Period A: SAR442970
Number analyzed (Participants) | 23 | 48
percentage of participants | 30.4 | 16.7

8. Secondary Outcome: Period A (DB Period): Percentage of Participants Who Achieved International Hidradenitis Suppurativa Severity Score System (IHS4)-55 at Week 16
Description: The IHS4 was a validated tool to assess HS severity. The determination of IHS4 required counting inflammatory nodules, abscesses and draining tunnels and multiplying each by a specific coefficient. IHS4 score was calculated as: (number of inflammatory nodules multiplied by 1) + (number of abscesses multiplied by 2) + (number of draining tunnels multiplied by 4). A categorial IHS4 score was derived from this weighted score with total score range: mild: (<=3), moderate: (4 to 10) and severe: (>=11); higher scores indicated worse outcomes. IHS4-55 was defined as a 55% reduction in IHS4 score from baseline. Baseline was defined as the last available value before the first dose of DB study drug.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Period A: Placebo | Period A: SAR442970
Number analyzed (Participants) | 23 | 48
percentage of participants | 34.8 | 64.6

9. Secondary Outcome: Period A (DB Period) + Period B (OLE Period): Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs) and Treatment-Emergent Adverse Events of Special Interest (TEAESIs)
Description: An AE as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE was defined as any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were AEs that developed, worsened or became serious during the TE period. An AESI was an AE (serious or non-serious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required.
Time Frame: Period A was assessed from first dose of study drug (Day 1 in Period A) up to last dose of study drug + 75 days, up to 192 days; Period B was assessed from first dose in Period B to last dose of study drug + 75 days, up to 168 days
Population: The safety population included for Period A: all randomized participants who had taken at least 1 dose of study drug during Period A, regardless of the amount of study drug administered and for Period B: all randomized participants who continued in Period B and who had taken at least 1 dose of study drug during Period B, regardless of the amount of study drug administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Period A: Placebo | Period A: SAR442970 | Period B: Placebo-SAR442970 | Period B: SAR442970-SAR442970
Number analyzed (Participants) | 28 | 58 | 26 | 51
Participants
  Any TEAEs | 15 | 45 | 14 | 30
  Any TESAEs | 0 | 0 | 0 | 0
  Any TEAESIs | 0 | 3 | 0 | 2

10. Secondary Outcome: Period A (DB Period): Percentage of Participants Who Achieved at Least 30% Reduction and at Least 1 Unit Reduction From Baseline in Weekly Average of Daily Hidradenitis Suppurativa Skin Pain Numeric Rating Scale (HS-Skin Pain NRS) at Week 16
Description: The HS-Skin Pain NRS was a unidimensional numeric rating scale (NRS) that allowed for rapid measure of skin pain that was administered multiple times with minimal administrative burden. The HS-Skin Pain NRS had a 24-hour recall period and was completed as a daily diary, ideally at the same time each day (evening) throughout the treatment period. Participants were asked to complete the HS-Skin Pain NRS for 7 consecutive days leading up to the baseline visit with a minimum of 4 completions in their daily diary. The HS-Skin Pain NRS was scored on a 0 to 10 scale; 0: no skin pain and 10: worst skin pain possible. Higher scores indicated worse outcomes. Baseline was defined as the last available value before the first dose of DB study drug.
Time Frame: Baseline (Day 1) and Week 16
Population: The biologic and small molecule immunosuppressive-naïve population included all randomized participants in the biologic and small molecule immunosuppressive-naïve subgroup who had taken at least 1 dose of study drug during Period A. Only those participants with Baseline NRS >=3 are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Period A: Placebo | Period A: SAR442970
Number analyzed (Participants) | 15 | 32
percentage of participants | 40.0 | 40.6

11. Secondary Outcome: Period A (DB Period) + Period B (OLE Period): Serum SAR442970 Concentrations
Description: Blood samples were collected at specified timepoints for assessment of serum SAR442970 concentrations.
Time Frame: Baseline (Day 1), Weeks 4, 8, 10, 12 and 16 (Period A); Weeks 18, 20 and 28 (Period B)
Population: The pharmacokinetic (PK) population included for Period A: all participants from the safety population of Period A with at least 1 post-Baseline PK result and for Period B: all participants from the safety population of Period B with at least 1 post-Baseline PK result. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Period A: SAR442970 | Period B: Placebo-SAR442970 | Period B: SAR442970-SAR442970
Number analyzed (Participants) | 58 | 25 | 48
nanogram per milliliter
  Baseline (Day 1): number analyzed (Participants) | 58 | 0 | 0
  Baseline (Day 1) | 0.00 (0.00) |  |
  Week 4: number analyzed (Participants) | 56 | 0 | 0
  Week 4 | 6451.21 (2252.03) |  |
  Week 8: number analyzed (Participants) | 53 | 0 | 0
  Week 8 | 7729.59 (2957.15) |  |
  Week 10: number analyzed (Participants) | 55 | 0 | 0
  Week 10 | 8091.69 (5141.56) |  |
  Week 12: number analyzed (Participants) | 53 | 0 | 0
  Week 12 | 9486.51 (8715.72) |  |
  Week 16: number analyzed (Participants) | 52 | 0 | 0
  Week 16 | 8844.81 (5908.33) |  |
  Week 18: number analyzed (Participants) | 0 | 23 | 48
  Week 18 |  | 4696.96 (1941.04) | 7996.88 (3716.46)
  Week 20: number analyzed (Participants) | 0 | 25 | 48
  Week 20 |  | 5693.20 (2223.45) | 8339.58 (4192.17)
  Week 28: number analyzed (Participants) | 0 | 23 | 43
  Week 28 |  | 7291.30 (3197.02) | 8513.07 (6868.14)

12. Secondary Outcome: Period B (OLE Period) + Period A+B (DB+OLE Period): Number of Participants With Anti-SAR442970 Antibody Response
Description: Serum samples were collected at specified timepoints for assessment of anti-SAR442970 antibody response. Treatment-emergent anti-drug antibody (ADA) were defined as participants with at least 1 treatment-induced/boosted ADA at any time after first study drug administration up to the last available ADA sample collection. Number of participants with treatment-emergent ADA response are presented.
Time Frame: Period B: Placebo-SAR442970 arm were assessed from first dose of study drug in Period B up to approximately 20 weeks. Period A+B: SAR442970-SAR442970 arm were assessed from first dose of study drug in Period A up to 36 weeks
Population: All participants from the ADA population, i.e., treated with SAR442970 with at least 1 post-baseline ADA result are included in Part B arm and in Parts A+B arm. The combined ADA analysis provided the accurate summary of all treatment-emergent ADA response in both treatment groups after the initiation of SAR443820.
Measure: Count of Participants; unit: Participants
Groups:
- Period A+B: SAR442970-SAR442970: Participants who received SAR442970 in Period A (DB period) received SAR442970 150 mg Q2W via SC injection from Week 16 to Week 28 in Period B (OLE period).
Arm/Group | Period B: Placebo-SAR442970 | Period A+B: SAR442970-SAR442970
Number analyzed (Participants) | 25 | 58
Participants | 18 | 45

ADVERSE EVENTS:
Time Frame: AEs and SAEs: Period A was assessed from first dose of study drug (Day 1 in Period A) up to last dose of study drug + 75 days, up to 192 days; Period B was assessed from first dose in Period B to last dose of study drug + 75 days, up to 168 days. All-cause mortality (deaths) were collected from the first dose of study drug to the end of follow-up for death for each participant, up to approximately 583 days.
Description: Analysis was performed on the safety population.
Arm/Group | Period A: Placebo | Period A: SAR442970 | Period B: Placebo-SAR442970 | Period B: SAR442970-SAR442970
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/58 | 0/26 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/58 | 0/26 | 0/51
Other Adverse Events (participants affected / at risk) | 11/28 | 32/58 | 6/26 | 16/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period A: Placebo (N=28) | Period A: SAR442970 (N=58) | Period B: Placebo-SAR442970 (N=26) | Period B: SAR442970-SAR442970 (N=51)
Nasopharyngitis (Infections and infestations) | 3 (3) | 11 (11) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 4 (4) | 2 (3) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 8 (16) | 2 (2) | 4 (5)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Injection Site Reaction (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 4 (4) | 7 (7) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT05849922/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT05849922/SAP_001.pdf